CLINICAL TRIAL: NCT04881760
Title: A Phase 2 Study of Once-Weekly LY3437943 Compared With Placebo in Participants Who Have Obesity or Are Overweight With Weight-Related Comorbidities
Brief Title: A Study of LY3437943 in Participants Who Have Obesity or Are Overweight
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18122; J1I-MC-GZBF (Other: Eli Lilly and Company)
Record Dates: First submitted 2021-05-10; First posted 2021-05-11 (Actual); Results first posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Obesity; Overweight
Keywords: Nutritional or Metabolism Disorder; Weight Loss; Overnutrition; Incretins; Hormones; Physiological Effects of Drugs
MeSH Terms: conditions — Obesity; Overweight; Metabolic Diseases; Weight Loss; Overnutrition | interventions — retatrutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Placebo (Placebo Comparator): Participants received placebo matched to LY3437943 administered as subcutaneous (SC) injection once-weekly (QW).
  Interventions: Drug: Placebo
- 1 milligram (mg) LY3437943 (Experimental): Participants received 1 mg LY3437943 administered as SC injection QW.
  Interventions: Drug: LY3437943
- 4 mg LY3437943 (2 mg) (Experimental): Participants received 2 mg LY3437943 starting dose followed by 4 mg LY3437943 administered as SC injection QW.
  Interventions: Drug: LY3437943
- 4 mg LY3437943 (Experimental): Participants received 4 mg LY3437943 administered as SC injection QW.
  Interventions: Drug: LY3437943
- 8 mg LY3437943 (2 mg) (Experimental): Participants received 2 mg LY3437943 starting dose followed by 4 mg LY3437943 and then 8 mg LY3437943 administered as SC injection QW.
  Interventions: Drug: LY3437943
- 8 mg LY3437943 (4 mg) (Experimental): Participants received 4 mg LY3437943 starting dose followed by 8 mg LY3437943 administered as SC injection QW.
  Interventions: Drug: LY3437943
- 12 mg LY3437943 (2 mg) (Experimental): Participants received 2 mg LY3437943 starting dose followed by 4 mg LY3437943, 8 mg LY3437943 and then 12 mg LY3437943 administered as SC injection QW.
  Interventions: Drug: LY3437943

INTERVENTIONS:
Drug: LY3437943 — Administered SC
  Arms: 1 milligram (mg) LY3437943; 12 mg LY3437943 (2 mg); 4 mg LY3437943; 4 mg LY3437943 (2 mg); 8 mg LY3437943 (2 mg); 8 mg LY3437943 (4 mg)
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
This is a study of LY3437943 in participants who have obesity or are overweight. The main purpose is to learn more about how LY3437943 affects body weight loss. The study will last about 18 months and may include up to 18 visits.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a Body Mass Index (BMI) ) ≥30 and ≤50 kilograms per square meter (kg/m²), or ≥27 kg/m² and <30 kg/m², with at least one of the following comorbidities: hypertension, dyslipidemia, cardiovascular disease
* Participants must be willing to learn how to self-inject study drug or receive an injection from a trained individual if visually impaired or with physical limitations, and follow study procedures for the duration of the study, including, but not limited to, follow lifestyle advice (for example, dietary changes and physical activity plan), maintain a study drug administration log, and complete required questionnaires

Exclusion Criteria:

* Participants must not have type 1 or type 2 diabetes mellitus
* Participants must not have had an increase or decrease in body weight > more than 5 kg (11 pounds) within the past 3 months
* Participants must not have had surgery for obesity or plan to have such surgery during the study
* Participants must not be using medications that promote weight loss or cause weight gain
* Participants must not drink excessive amounts of alcohol (more than 14 units a week for women or more than 21 units a week for men)
* Participants must not have used marijuana within the last 3 months.
* Participants must not have heart attack, stroke, or hospitalization for congestive heart failure in the past 3 months
* Participants must not have active cancer within the last 5 years
* Participants must not have uncontrolled high blood pressure
* Participants must not have liver disease other than non-alcoholic fatty liver disease
* Participants must not have renal impairment with estimated glomerular filtration rate (eGFR) <45 mL/min/1.73 m2
* Participants must not have a history of acute or chronic pancreatitis symptomatic gallbladder disease or documented human immunodeficiency virus infection
* Participants must not have a major problem with depression or other mental illness within the last 2 years
* Participants must not have family or personal history of multiple endocrine neoplasia type 2 or medullary thyroid carcinoma (family is defined as a first degree relative)
* Female participants must not be pregnant, breast-feeding, or intend to become pregnant or of childbearing potential and not using adequate contraceptive method (adequate contraceptive measures as required by local regulation or practice)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (28):
- United States (25):
  - Perseverance Research Center, Scottsdale, Arizona
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Valley Research, Fresno, California
  - Velocity Clinical Research, Huntington Park, Huntington Park, California
  - Velocity Clinical Research, Huntington Park, Los Angeles, California
  - Southern California Dermatology, Inc., Santa Ana, California
  - Coastal Metabolic Research Centre, Ventura, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - East Coast Institute for Research, LLC, Jacksonville, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Encore Medical Research - Weston, Weston, Florida
  - Springfield Diabetes & Endocrine Center, Springfield, Illinois
  - Cotton O'Neil Diabetes and Endocrinology Center, Topeka, Kansas
  - Tandem Clinical Research,LLC, Marrero, Louisiana
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Amici Clinical Research LLC, Raritan, New Jersey
  - Intend Research, LLC, Norman, Oklahoma
  - Allegheny Endocrinology Associates, Pittsburgh, Pennsylvania
  - New Phase Research and Development, Knoxville, Tennessee
  - Texas Diabetes & Endocrinology, P.A., Austin, Texas
  - Dallas Diabetes Research Center, Dallas, Texas
  - Juno Research, Houston, Texas
  - Endocrine Ips, Pllc, Houston, Texas
  - Southern Endocrinology Associates, Mesquite, Texas
  - Rainier Clinical Research Center, Renton, Washington
- Puerto Rico (3):
  - Private Practice - Dr. Paola Mansilla-Letelier, Guaynabo
  - GCM Medical Group, PSC - Hato Rey Site, San Juan
  - San Juan City Hospital, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Sanyal AJ, Kaplan LM, Frias JP, Brouwers B, Wu Q, Thomas MK, Harris C, Schloot NC, Du Y, Mather KJ, Haupt A, Hartman ML. Triple hormone receptor agonist retatrutide for metabolic dysfunction-associated steatotic liver disease: a randomized phase 2a trial. Nat Med. 2024 Jul;30(7):2037-2048. doi: 10.1038/s41591-024-03018-2. Epub 2024 Jun 10. PMID 38858523
- [Derived] Jastreboff AM, Kaplan LM, Frias JP, Wu Q, Du Y, Gurbuz S, Coskun T, Haupt A, Milicevic Z, Hartman ML; Retatrutide Phase 2 Obesity Trial Investigators. Triple-Hormone-Receptor Agonist Retatrutide for Obesity - A Phase 2 Trial. N Engl J Med. 2023 Aug 10;389(6):514-526. doi: 10.1056/NEJMoa2301972. Epub 2023 Jun 26. PMID 37366315
- See also: A Study of LY3437943 in Participants Who Have Obesity or Are Overweight — https://trials.lillytrialguide.com/en-US/trial/36s0UdwlFjVCXwfbif2fkc

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Four maintenance doses of LY3437943 were evaluated in the trial: 1, 4, 8, and 12 milligrams (mg). Dose escalation to improve gastrointestinal (GI) tolerability occured in certain treatment groups up to Week 12 by increasing the volume of administered study drug (or placebo) during the 48-week double-blind, placebo-controlled treatment period.
Groups:
- 1 mg LY3437943: Participants received 1 mg LY3437943 administered as SC injection QW.
Period: Overall Study
Arm/Group | Placebo | 1 mg LY3437943 | 4 mg LY3437943 (2 mg) | 4 mg LY3437943 | 8 mg LY3437943 (2 mg) | 8 mg LY3437943 (4 mg) | 12 mg LY3437943 (2 mg)
Started | 70 | 69 | 33 | 34 | 35 | 35 | 62
Received at Least One Dose of Study Drug | 70 | 69 | 33 | 33 | 35 | 35 | 62
Completed | 50 | 60 | 26 | 26 | 30 | 29 | 54
Not Completed | 20 | 9 | 7 | 8 | 5 | 6 | 8
Not completed — Adverse Event | 0 | 1 | 1 | 0 | 1 | 1 | 2
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 5 | 7 | 5 | 1 | 2 | 4 | 4
Not completed — Withdrawal by Subject | 13 | 1 | 1 | 4 | 2 | 1 | 2
Not completed — Randomized but Never Treated | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Inadvertent Enrollment | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Site Closure | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Placebo: Participants received placebo matched to LY3437943 administered as SC injection QW.
- 8 mg LY343794 (4 mg): Participants received 4 mg LY3437943 starting dose followed by 8 mg LY3437943 administered as SC injection QW.
- Total: Total of all reporting groups
Arm/Group | Placebo | 1 mg LY3437943 | 4 mg LY3437943 (2 mg) | 4 mg LY3437943 | 8 mg LY3437943 (2 mg) | 8 mg LY343794 (4 mg) | 12 mg LY3437943 (2 mg) | Total
Number analyzed (Participants) | 70 | 69 | 33 | 34 | 35 | 35 | 62 | 338
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.00 (12.54) | 50.60 (13.30) | 50.80 (11.88) | 46.80 (14.10) | 46.10 (13.52) | 48.70 (11.14) | 45.80 (12.18) | 48.20 (12.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 33 | 16 | 16 | 17 | 17 | 30 | 163
  Male | 36 | 36 | 17 | 18 | 18 | 18 | 32 | 175
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 23 | 9 | 14 | 15 | 12 | 22 | 117
  Not Hispanic or Latino | 47 | 46 | 24 | 20 | 20 | 23 | 40 | 220
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
  Asian | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 8 | 6 | 4 | 2 | 4 | 1 | 2 | 27
  White | 59 | 61 | 29 | 30 | 30 | 33 | 56 | 298
  More than one race | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 5
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 70 | 69 | 33 | 34 | 35 | 35 | 62 | 338
Baseline Body Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 109.21 (20.88) | 106.36 (19.84) | 108.04 (26.31) | 107.01 (21.29) | 106.50 (21.55) | 108.63 (20.88) | 107.97 (21.69) | 107.73 (21.35)
Baseline Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per meter squared (kg/m^2)] | 37.31 (5.90) | 37.49 (5.85) | 37.27 (5.87) | 37.39 (4.66) | 37.37 (6.04) | 36.96 (5.49) | 37.42 (5.98) | 37.34 (5.71)

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change From Baseline in Body Weight
Description: Least squares (LS) means were calculated using a mixed-effects model for repeated measures (MMRM) for post-baseline measures: Variable = Treatment*Time + Baseline BMI (< 36kg/m2 vs. >=36 kg/m2)*Time + Sex (Female vs. Male)*Time + Baseline*Time.
Time Frame: Baseline, Week 24
Population: All randomized participants who had baseline and at least one post-baseline body weight value, excluding participants discontinuing study drug due to inadvertent enrollment and data after discontinuation of study drug.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | 1 mg LY3437943 | 4 mg LY3437943 (2 mg) | 4 mg LY3437943 | 8 mg LY3437943 (2 mg) | 8 mg LY3437943 (4 mg) | 12 mg LY3437943 (2 mg)
Number analyzed (Participants) | 68 | 69 | 33 | 33 | 35 | 35 | 62
percent change | -1.55 (0.54) | -7.18 (0.67) | -12.00 (0.71) | -13.80 (0.97) | -16.64 (0.74) | -18.26 (0.95) | -17.39 (0.69)
Statistical Analysis 1: Comparison: Placebo vs 1 mg LY3437943; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -5.64, 95% CI 2-sided [-7.34 to -3.94]
Statistical Analysis 2: Comparison: Placebo vs 4 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -10.45, 95% CI 2-sided [-12.21 to -8.70]
Statistical Analysis 3: Comparison: Placebo vs 4 mg LY3437943; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -12.25, 95% CI 2-sided [-14.42 to -10.08]
Statistical Analysis 4: Comparison: Placebo vs 8 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -15.10, 95% CI 2-sided [-16.90 to -13.30]
Statistical Analysis 5: Comparison: Placebo vs 8 mg LY3437943 (4 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -16.72, 95% CI 2-sided [-18.86 to -14.58]
Statistical Analysis 6: Comparison: Placebo vs 12 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -15.85, 95% CI 2-sided [-17.57 to -14.13]

2. Secondary Outcome: Mean Percent Change From Baseline in Body Weight
Description: LS means were calculated using a MMRM model for post-baseline measures: Variable = Treatment*Time + Baseline BMI (< 36kg/m2 vs. >=36 kg/m2)*Time + Sex (Female vs. Male)*Time + Baseline*Time.
Time Frame: Baseline, Week 48
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | 1 mg LY3437943 | 4 mg LY3437943 (2 mg) | 4 mg LY3437943 | 8 mg LY3437943 (2 mg) | 8 mg LY3437943 (4 mg) | 12 mg LY3437943 (2 mg)
Number analyzed (Participants) | 68 | 69 | 33 | 33 | 35 | 35 | 62
percent change | -2.11 (0.73) | -8.67 (0.95) | -16.32 (1.58) | -17.83 (1.53) | -21.72 (1.41) | -23.88 (1.51) | -24.22 (1.24)
Statistical Analysis 1: Comparison: Placebo vs 1 mg LY3437943; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -6.57, 95% CI 2-sided [-8.94 to -4.20]
Statistical Analysis 2: Comparison: Placebo vs 4 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -14.21, 95% CI 2-sided [-17.64 to -10.78]
Statistical Analysis 3: Comparison: Placebo vs 4 mg LY3437943; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -15.72, 95% CI 2-sided [-19.05 to -12.40]
Statistical Analysis 4: Comparison: Placebo vs 8 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -19.62, 95% CI 2-sided [-22.73 to -16.51]
Statistical Analysis 5: Comparison: Placebo vs 8 mg LY3437943 (4 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -21.78, 95% CI 2-sided [-25.05 to -18.51]
Statistical Analysis 6: Comparison: Placebo vs 12 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -22.11, 95% CI 2-sided [-24.92 to -19.31]

3. Secondary Outcome: Percentage of Participants Who Achieve ≥ 5% Body Weight Reduction
Description: Percentage of participants who achieve ≥ 5% body weight reduction in LY3437943 relative to placebo. Estimated percentage was determined by logistic regression model with an intercept term, treatment group, baseline BMI stratum [<36 kilograms per square meter (kg/m2), ≥36 kg/m2] and sex [female, male] as fixed effects, and baseline body weight as a covariate.
Time Frame: Week 24
Population: All randomized participants who had baseline and at least one post-baseline value for ≥ 5% body weight reduction excluding participants discontinuing study drug due to inadvertent enrollment and data after discontinuation of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 1 mg LY3437943 | 4 mg LY3437943 (2 mg) | 4 mg LY3437943 | 8 mg LY3437943 (2 mg) | 8 mg LY3437943 (4 mg) | 12 mg LY3437943 (2 mg)
Number analyzed (Participants) | 68 | 69 | 33 | 33 | 35 | 35 | 62
percentage of participants | 26 | 59 | 87 | 94 | 100 | 100 | 97
Statistical Analysis 1: Comparison: Placebo vs 1 mg LY3437943; Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 33, 95% CI 2-sided [17 to 49]
Statistical Analysis 2: Comparison: Placebo vs 4 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 61, 95% CI 2-sided [45 to 77]
Statistical Analysis 3: Comparison: Placebo vs 4 mg LY3437943; Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 68, 95% CI 2-sided [54 to 81]
Statistical Analysis 4: Comparison: Placebo vs 8 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 74, 95% CI 2-sided [63 to 85]
Statistical Analysis 5: Comparison: Placebo vs 8 mg LY3437943 (4 mg); Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 74, 95% CI 2-sided [63 to 85]
Statistical Analysis 6: Comparison: Placebo vs 12 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 71, 95% CI 2-sided [59 to 82]

4. Secondary Outcome: Percentage of Participants Who Achieve ≥ 5% Body Weight Reduction
Description: Percentage of participants who achieve ≥ 5% body weight reduction in LY3437943 relative to placebo. Estimated percentage was determined by logistic regression model with an intercept term, treatment group, baseline BMI stratum [<36 kg/m2, ≥36 kg/m2] and sex [female, male] as fixed effects, and baseline body weight as a covariate.
Time Frame: Week 48
Population: All randomized participants who had baseline and at least one post-baseline value for ≥ 5% body weight reduction, excluding participants discontinuing study drug due to inadvertent enrollment and data after discontinuation of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 1 mg LY3437943 | 4 mg LY3437943 (2 mg) | 4 mg LY3437943 | 8 mg LY3437943 (2 mg) | 8 mg LY3437943 (4 mg) | 12 mg LY3437943 (2 mg)
Number analyzed (Participants) | 68 | 69 | 33 | 33 | 35 | 35 | 62
percentage of participants | 27 | 64 | 87 | 97 | 100 | 100 | 100
Statistical Analysis 1: Comparison: Placebo vs 1 mg LY3437943; Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 37, 95% CI 2-sided [20 to 54]
Statistical Analysis 2: Comparison: Placebo vs 4 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 60, 95% CI 2-sided [44 to 76]
Statistical Analysis 3: Comparison: Placebo vs 4 mg LY3437943; Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 70, 95% CI 2-sided [57 to 83]
Statistical Analysis 4: Comparison: Placebo vs 8 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 73, 95% CI 2-sided [62 to 84]
Statistical Analysis 5: Comparison: Placebo vs 8 mg LY3437943 (4 mg); Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 73, 95% CI 2-sided [62 to 84]
Statistical Analysis 6: Comparison: Placebo vs 12 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 73, 95% CI 2-sided [67 to 84]

5. Secondary Outcome: Percentage of Participants Who Achieve ≥ 10% Body Weight Reduction
Description: Percentage of participants who achieve ≥ 10% body weight reduction in LY3437943 relative to placebo. Estimated percentage was determined by logistic regression model with an intercept term, treatment group, baseline BMI stratum [<36 kg/m2, ≥36 kg/m2] and sex [female, male] as fixed effects, and baseline body weight as a covariate.
Time Frame: Week 24
Population: All randomized participants who had baseline and at least one post-baseline value for ≥ 10% body weight reduction, excluding participants discontinuing study drug due to inadvertent enrollment and data after discontinuation of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 1 mg LY3437943 | 4 mg LY3437943 (2 mg) | 4 mg LY3437943 | 8 mg LY3437943 (2 mg) | 8 mg LY3437943 (4 mg) | 12 mg LY3437943 (2 mg)
Number analyzed (Participants) | 68 | 69 | 33 | 33 | 35 | 35 | 62
percentage of participants | 3 | 25 | 59 | 72 | 83 | 94 | 90
Statistical Analysis 1: Comparison: Placebo vs 1 mg LY3437943; Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 22, 95% CI 2-sided [11 to 33]
Statistical Analysis 2: Comparison: Placebo vs 4 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 56, 95% CI 2-sided [38 to 73]
Statistical Analysis 3: Comparison: Placebo vs 4 mg LY3437943; Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 69, 95% CI 2-sided [53 to 85]
Statistical Analysis 4: Comparison: Placebo vs 8 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 80, 95% CI 2-sided [66 to 93]
Statistical Analysis 5: Comparison: Placebo vs 8 mg LY3437943 (4 mg); Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 91, 95% CI 2-sided [83 to 100]
Statistical Analysis 6: Comparison: Placebo vs 12 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 87, 95% CI 2-sided [78 to 96]

6. Secondary Outcome: Percentage of Participants Who Achieve ≥ 10% Body Weight Reduction
Description: as for outcome 5
Time Frame: Week 48
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 1 mg LY3437943 | 4 mg LY3437943 (2 mg) | 4 mg LY3437943 | 8 mg LY3437943 (2 mg) | 8 mg LY3437943 (4 mg) | 12 mg LY3437943 (2 mg)
Number analyzed (Participants) | 68 | 69 | 33 | 33 | 35 | 35 | 62
percentage of participants | 9 | 27 | 73 | 76 | 90 | 91 | 93
Statistical Analysis 1: Comparison: Placebo vs 1 mg LY3437943; Test type: Superiority; p = 0.008, Regression, Logistic; Risk Difference (RD) = 18, 95% CI 2-sided [5 to 31]
Statistical Analysis 2: Comparison: Placebo vs 4 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 64, 95% CI 2-sided [48 to 81]
Statistical Analysis 3: Comparison: Placebo vs 4 mg LY3437943; Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 67, 95% CI 2-sided [51 to 84]
Statistical Analysis 4: Comparison: Placebo vs 8 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 81, 95% CI 2-sided [69 to 94]
Statistical Analysis 5: Comparison: Placebo vs 8 mg LY3437943 (4 mg); Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 82, 95% CI 2-sided [71 to 94]
Statistical Analysis 6: Comparison: Placebo vs 12 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 84, 95% CI 2-sided [74 to 94]

7. Secondary Outcome: Percentage of Participants Who Achieve ≥ 15% Body Weight Reduction
Description: Percentage of participants who achieve ≥ 15% body weight reduction in LY3437943 relative to placebo. Estimated percentage was determined by logistic regression model with an intercept term, treatment group, baseline BMI stratum [<36 kg/m2, ≥36 kg/m2] and sex [female, male] as fixed effects, and baseline body weight as a covariate.
Time Frame: Week 24
Population: All randomized participants who had baseline and at least one post-baseline value for ≥ 15% body weight reduction, excluding participants discontinuing study drug due to inadvertent enrollment and data after discontinuation of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 1 mg LY3437943 | 4 mg LY3437943 (2 mg) | 4 mg LY3437943 | 8 mg LY3437943 (2 mg) | 8 mg LY3437943 (4 mg) | 12 mg LY3437943 (2 mg)
Number analyzed (Participants) | 68 | 69 | 33 | 33 | 35 | 35 | 62
percentage of participants | 1 | 10 | 29 | 44 | 51 | 68 | 70
Statistical Analysis 1: Comparison: Placebo vs 1 mg LY3437943; Test type: Superiority; p = 0.029, Regression, Logistic; Risk Difference (RD) = 9, 95% CI 2-sided [1 to 17]
Statistical Analysis 2: Comparison: Placebo vs 4 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 27, 95% CI 2-sided [11 to 43]
Statistical Analysis 3: Comparison: Placebo vs 4 mg LY3437943; Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 43, 95% CI 2-sided [26 to 60]
Statistical Analysis 4: Comparison: Placebo vs 8 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 49, 95% CI 2-sided [33 to 66]
Statistical Analysis 5: Comparison: Placebo vs 8 mg LY3437943 (4 mg); Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 67, 95% CI 2-sided [51 to 83]
Statistical Analysis 6: Comparison: Placebo vs 12 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 68, 95% CI 2-sided [56 to 80]

8. Secondary Outcome: Percentage of Participants Who Achieve ≥ 15% Body Weight Reduction
Description: as for outcome 7
Time Frame: Week 48
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 1 mg LY3437943 | 4 mg LY3437943 (2 mg) | 4 mg LY3437943 | 8 mg LY3437943 (2 mg) | 8 mg LY3437943 (4 mg) | 12 mg LY3437943 (2 mg)
Number analyzed (Participants) | 68 | 69 | 33 | 33 | 35 | 35 | 62
percentage of participants | 2 | 16 | 55 | 64 | 73 | 77 | 83
Statistical Analysis 1: Comparison: Placebo vs 1 mg LY3437943; Test type: Superiority; p = 0.002, Regression, Logistic; Risk Difference (RD) = 15, 95% CI 2-sided [6 to 24]
Statistical Analysis 2: Comparison: Placebo vs 4 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 53, 95% CI 2-sided [36 to 70]
Statistical Analysis 3: Comparison: Placebo vs 4 mg LY3437943; Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 63, 95% CI 2-sided [47 to 79]
Statistical Analysis 4: Comparison: Placebo vs 8 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 71, 95% CI 2-sided [55 to 87]
Statistical Analysis 5: Comparison: Placebo vs 8 mg LY3437943 (4 mg); Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 75, 95% CI 2-sided [62 to 89]
Statistical Analysis 6: Comparison: Placebo vs 12 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 82, 95% CI 2-sided [71 to 92]

9. Secondary Outcome: Mean Change From Baseline in Body Weight
Description: as for outcome 2
Time Frame: Baseline, Week 24
Population: All randomized participants who had baseline and at least one post-baseline value for body weight, excluding participants discontinuing study drug due to inadvertent enrollment and data after discontinuation of study drug.
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | Placebo | 1 mg LY3437943 | 4 mg LY3437943 (2 mg) | 4 mg LY3437943 | 8 mg LY3437943 (2 mg) | 8 mg LY3437943 (4 mg) | 12 mg LY3437943 (2 mg)
Number analyzed (Participants) | 68 | 69 | 33 | 33 | 35 | 35 | 62
kilograms (kg) | -1.27 (0.63) | -7.72 (0.73) | -12.59 (0.81) | -14.79 (1.09) | -17.70 (0.79) | -19.75 (1.08) | -18.53 (0.71)
Statistical Analysis 1: Comparison: Placebo vs 1 mg LY3437943; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -6.46, 95% CI 2-sided [-8.36 to -4.56]
Statistical Analysis 2: Comparison: Placebo vs 4 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -11.32, 95% CI 2-sided [-13.34 to -9.30]
Statistical Analysis 3: Comparison: Placebo vs 4 mg LY3437943; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -13.52, 95% CI 2-sided [-15.99 to -11.05]
Statistical Analysis 4: Comparison: Placebo vs 8 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -16.43, 95% CI 2-sided [-18.41 to -14.45]
Statistical Analysis 5: Comparison: Placebo vs 8 mg LY3437943 (4 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -18.48, 95% CI 2-sided [-20.93 to -16.04]
Statistical Analysis 6: Comparison: Placebo vs 12 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -17.26, 95% CI 2-sided [-19.11 to -15.40]

10. Secondary Outcome: Mean Change From Baseline in Body Weight
Description: as for outcome 2
Time Frame: Baseline, Week 48
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Placebo | 1 mg LY3437943 | 4 mg LY3437943 (2 mg) | 4 mg LY3437943 | 8 mg LY3437943 (2 mg) | 8 mg LY3437943 (4 mg) | 12 mg LY3437943 (2 mg)
Number analyzed (Participants) | 68 | 69 | 33 | 33 | 35 | 35 | 62
kg | -1.84 (0.83) | -9.37 (1.06) | -17.32 (1.78) | -19.13 (1.80) | -23.52 (1.61) | -25.88 (1.68) | -26.17 (1.33)
Statistical Analysis 1: Comparison: Placebo vs 1 mg LY3437943; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -7.53, 95% CI 2-sided [-10.18 to -4.88]
Statistical Analysis 2: Comparison: Placebo vs 4 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -15.48, 95% CI 2-sided [-19.35 to -11.60]
Statistical Analysis 3: Comparison: Placebo vs 4 mg LY3437943; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -17.29, 95% CI 2-sided [-21.19 to -13.39]
Statistical Analysis 4: Comparison: Placebo vs 8 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -21.69, 95% CI 2-sided [-25.25 to -18.12]
Statistical Analysis 5: Comparison: Placebo vs 8 mg LY3437943 (4 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -24.04, 95% CI 2-sided [-27.72 to -20.36]
Statistical Analysis 6: Comparison: Placebo vs 12 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -24.34, 95% CI 2-sided [-27.40 to -21.27]

11. Secondary Outcome: Mean Change From Baseline in BMI
Description: as for outcome 2
Time Frame: Baseline, Week 24
Population: All randomized participants who had baseline and at least one post-baseline BMI value, excluding participants discontinuing study drug due to inadvertent enrollment and data after discontinuation of study drug.
Measure: Least Squares Mean (Standard Error); unit: kg/m^2
Arm/Group | Placebo | 1 mg LY3437943 | 4 mg LY3437943 (2 mg) | 4 mg LY3437943 | 8 mg LY3437943 (2 mg) | 8 mg LY3437943 (4 mg) | 12 mg LY3437943 (2 mg)
Number analyzed (Participants) | 68 | 69 | 33 | 33 | 35 | 35 | 62
kg/m^2 | -0.49 (0.21) | -2.64 (0.26) | -4.47 (0.28) | -5.13 (0.36) | -6.15 (0.27) | -6.84 (0.36) | -6.44 (0.25)
Statistical Analysis 1: Comparison: Placebo vs 1 mg LY3437943; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -2.15, 95% CI 2-sided [-2.80 to -1.50]
Statistical Analysis 2: Comparison: Placebo vs 4 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -3.98, 95% CI 2-sided [-4.66 to -3.29]
Statistical Analysis 3: Comparison: Placebo vs 4 mg LY3437943; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -4.64, 95% CI 2-sided [-5.46 to -3.82]
Statistical Analysis 4: Comparison: Placebo vs 8 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -5.66, 95% CI 2-sided [-6.34 to -4.99]
Statistical Analysis 5: Comparison: Placebo vs 8 mg LY3437943 (4 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -6.35, 95% CI 2-sided [-7.17 to -5.53]
Statistical Analysis 6: Comparison: Placebo vs 12 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -5.95, 95% CI 2-sided [-6.59 to -5.32]

12. Secondary Outcome: Mean Change From Baseline in BMI
Description: as for outcome 2
Time Frame: Baseline, Week 48
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: kg/m^2
Arm/Group | Placebo | 1 mg LY3437943 | 4 mg LY3437943 (2 mg) | 4 mg LY3437943 | 8 mg LY3437943 (2 mg) | 8 mg LY3437943 (4 mg) | 12 mg LY3437943 (2 mg)
Number analyzed (Participants) | 68 | 69 | 33 | 33 | 35 | 35 | 62
kg/m^2 | -0.72 (0.29) | -3.22 (0.37) | -6.14 (0.65) | -6.67 (0.59) | -8.12 (0.55) | -9.02 (0.57) | -9.14 (0.46)
Statistical Analysis 1: Comparison: Placebo vs 1 mg LY3437943; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -2.50, 95% CI 2-sided [-3.42 to -1.57]
Statistical Analysis 2: Comparison: Placebo vs 4 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -5.42, 95% CI 2-sided [-6.81 to -4.03]
Statistical Analysis 3: Comparison: Placebo vs 4 mg LY3437943; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -5.95, 95% CI 2-sided [-7.23 to -4.67]
Statistical Analysis 4: Comparison: Placebo vs 8 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -7.40, 95% CI 2-sided [-8.62 to -6.18]
Statistical Analysis 5: Comparison: Placebo vs 8 mg LY3437943 (4 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -8.30, 95% CI 2-sided [-9.55 to -7.05]
Statistical Analysis 6: Comparison: Placebo vs 12 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -8.42, 95% CI 2-sided [-9.49 to -7.35]

13. Secondary Outcome: Mean Change From Baseline in Waist Circumference
Description: as for outcome 2
Time Frame: Baseline, Week 24
Population: All randomized participants who had baseline and at least one post-baseline waist circumference value, excluding participants discontinuing study drug due to inadvertent enrollment and data after discontinuation of study drug.
Measure: Least Squares Mean (Standard Error); unit: centimeters (cm)
Arm/Group | Placebo | 1 mg LY3437943 | 4 mg LY3437943 (2 mg) | 4 mg LY3437943 | 8 mg LY3437943 (2 mg) | 8 mg LY3437943 (4 mg) | 12 mg LY3437943 (2 mg)
Number analyzed (Participants) | 67 | 69 | 32 | 33 | 35 | 35 | 62
centimeters (cm) | -2.60 (0.80) | -5.43 (0.94) | -10.33 (1.05) | -12.55 (1.00) | -13.74 (1.04) | -14.99 (0.98) | -14.33 (0.86)
Statistical Analysis 1: Comparison: Placebo vs 1 mg LY3437943; Test type: Superiority; p = 0.022, Mixed Models Analysis; LS Mean difference (Final Values) = -2.82, 95% CI 2-sided [-5.23 to -0.41]
Statistical Analysis 2: Comparison: Placebo vs 4 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -7.73, 95% CI 2-sided [-10.32 to -5.13]
Statistical Analysis 3: Comparison: Placebo vs 4 mg LY3437943; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -9.95, 95% CI 2-sided [-12.47 to -7.43]
Statistical Analysis 4: Comparison: Placebo vs 8 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -11.14, 95% CI 2-sided [-13.72 to -8.56]
Statistical Analysis 5: Comparison: Placebo vs 8 mg LY3437943 (4 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -12.38, 95% CI 2-sided [-14.87 to -9.90]
Statistical Analysis 6: Comparison: Placebo vs 12 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -11.73, 95% CI 2-sided [-14.04 to -9.43]

14. Secondary Outcome: Mean Change From Baseline in Waist Circumference
Description: as for outcome 2
Time Frame: Baseline, Week 48
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | Placebo | 1 mg LY3437943 | 4 mg LY3437943 (2 mg) | 4 mg LY3437943 | 8 mg LY3437943 (2 mg) | 8 mg LY3437943 (4 mg) | 12 mg LY3437943 (2 mg)
Number analyzed (Participants) | 67 | 69 | 32 | 33 | 35 | 35 | 62
cm | -2.64 (0.99) | -6.49 (1.12) | -14.58 (1.56) | -14.87 (1.73) | -18.53 (1.46) | -18.50 (1.52) | -19.60 (1.29)
Statistical Analysis 1: Comparison: Placebo vs 1 mg LY3437943; Test type: Superiority; p = 0.010, Mixed Models Analysis; LS Mean difference (Final Values) = -3.84, 95% CI 2-sided [-6.77 to -0.91]
Statistical Analysis 2: Comparison: Placebo vs 4 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -11.94, 95% CI 2-sided [-15.54 to -8.33]
Statistical Analysis 3: Comparison: Placebo vs 4 mg LY3437943; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -12.22, 95% CI 2-sided [-16.11 to -8.33]
Statistical Analysis 4: Comparison: Placebo vs 8 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -15.88, 95% CI 2-sided [-19.33 to -12.43]
Statistical Analysis 5: Comparison: Placebo vs 8 mg LY3437943 (4 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -15.85, 95% CI 2-sided [-19.39 to -12.31]
Statistical Analysis 6: Comparison: Placebo vs 12 mg LY3437943 (2 mg); Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -16.95, 95% CI 2-sided [-20.13 to -13.78]

ADVERSE EVENTS:
Time Frame: Baseline Through End of Safety Follow-up (Up to 52 Weeks)
Description: All randomized participants who received at least one dose of study drug, regardless of adherence to study drug. Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly. Frequency threshold for reporting other (not including serious) adverse event is greater than or equal to (≥) 5% in any of the treatment groups.
Groups:
- 8 mg LY3437943 (2 mg): Participants received 2 mg LY343794 starting dose followed by 4 mg LY3437943 and then 8 mg LY3437943 administered as SC injection QW.
Arm/Group | Placebo | 1 mg LY3437943 | 4 mg LY3437943 (2 mg) | 4 mg LY3437943 | 8 mg LY3437943 (2 mg) | 8 mg LY3437943 (4 mg) | 12 mg LY3437943 (2 mg)
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/69 | 0/33 | 1/33 | 0/35 | 0/35 | 0/62
Serious Adverse Events (participants affected / at risk) | 3/70 | 3/69 | 0/33 | 2/33 | 1/35 | 2/35 | 2/62
Other Adverse Events (participants affected / at risk) | 40/70 | 46/69 | 22/33 | 24/33 | 26/35 | 31/35 | 52/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=70) | 1 mg LY3437943 (N=69) | 4 mg LY3437943 (2 mg) (N=33) | 4 mg LY3437943 (N=33) | 8 mg LY3437943 (2 mg) (N=35) | 8 mg LY3437943 (4 mg) (N=35) | 12 mg LY3437943 (2 mg) (N=62)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drowning (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood calcitonin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=70) | 1 mg LY3437943 (N=69) | 4 mg LY3437943 (2 mg) (N=33) | 4 mg LY3437943 (N=33) | 8 mg LY3437943 (2 mg) (N=35) | 8 mg LY3437943 (4 mg) (N=35) | 12 mg LY3437943 (2 mg) (N=62)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 5 (6)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 3 (4) | 2 (2) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (3) | 5 (7) | 5 (6) | 2 (3) | 4 (5) | 4 (4) | 10 (13)
Diarrhoea (Gastrointestinal disorders) | 8 (9) | 6 (8) | 4 (5) | 4 (5) | 7 (11) | 7 (9) | 9 (17)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 2 (3) | 2 (2) | 5 (7)
Faeces hard (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 3 (3) | 0 (0) | 4 (8)
Nausea (Gastrointestinal disorders) | 8 (8) | 10 (12) | 6 (9) | 12 (21) | 6 (9) | 21 (33) | 28 (63)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 4 (6) | 4 (5) | 2 (3) | 9 (9) | 12 (21)
Early satiety (General disorders) | 4 (4) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 6 (6)
Fatigue (General disorders) | 3 (4) | 3 (4) | 4 (4) | 2 (2) | 1 (1) | 3 (3) | 6 (6)
Covid-19 (Infections and infestations) | 14 (14) | 13 (13) | 4 (4) | 6 (6) | 6 (6) | 11 (11) | 15 (15)
Nasopharyngitis (Infections and infestations) | 3 (3) | 6 (6) | 0 (0) | 2 (2) | 3 (4) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 4 (5) | 2 (2) | 1 (1) | 1 (3) | 1 (2) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 1 (2) | 0 (0) | 2 (3) | 2 (3)
Vaginal infection (Infections and infestations) | 0/34 (0) | 0/33 (0) | 0/16 (0) | 1/15 (1) | 0/17 (0) | 0/17 (0) | 0/30 (0)
Amylase increased (Investigations) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 5 (5) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Lipase increased (Investigations) | 2 (2) | 2 (2) | 3 (3) | 2 (2) | 1 (1) | 2 (2) | 5 (5)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6) | 9 (10) | 6 (6) | 8 (8) | 4 (5) | 11 (12) | 18 (19)
Allodynia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 5 (9)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 4 (6)
Hyperaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 0/36 (0) | 2/36 (2) | 0/17 (0) | 0/18 (0) | 0/18 (0) | 0/18 (0) | 0/32 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 2 (2)
Sensitive skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Hypertension (Vascular disorders) | 2 (2) | 6 (6) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 4 (4)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-08-29): https://cdn.clinicaltrials.gov/large-docs/60/NCT04881760/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-15): https://cdn.clinicaltrials.gov/large-docs/60/NCT04881760/SAP_001.pdf